CLINICAL TRIAL: NCT06076369
Title: Differentiation of Tubular Adenoma IIIL Duct Opening and Colonic Innominate Groove Under EC Endoscopy
Brief Title: Differentiation of Tubular Adenoma and Colonic Innominate Groove Under EC Endoscopy
Status: Recruiting | Type: Observational
Sponsor: Jilin University (Other)
Responsible Party: Principal Investigator, Dong Yang, Assisted Investigator, Jilin University
Other Study IDs: 130025
Record Dates: First submitted 2023-08-23; First posted 2023-10-10 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: Endocytoscopy
Keywords: tubular adenoma; IIIL duct opening; colonic innominate groove

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- The tubular adenoma group: The anatomical site was determined, and the size and morphology of the polyps were observed. The classification of the microvascular ECV of the polyps and its adjacent normal mucosal microvascular ECV (white light+NBI) was observed, and methylene blue staining was used to approach and magnify the glandular duct opening to observe the IIIL type (pit pattern). Magnified to the maximum magnification of EC endoscopy to the clearest cell level (approximately 520 times), and observed the morphology of the opening of the IIIL type glandular duct and the opening of the colonic innominate groove, including the morphology of cell cytoplasm and nucleus, proportion of opening length to field of view (more than 1 field of view is calculated as 1.0), and ratio of maximum to minimum opening diameter; Distribution characteristics of glandular duct openings.
  Interventions: Procedure: The tubular adenoma group
- the colonic innominate groove group: The methylene blue staining area of the normal mucosa adjacent to the polyp was observed to identify the colonic innominate groove.Magnified to the maximum magnification of EC endoscopy to the clearest cell level (approximately 520 times), and observed the morphology of the opening of the IIIL type glandular duct and the opening of the colonic innominate groove, including the morphology of cell cytoplasm and nucleus, proportion of opening length to field of view (more than 1 field of view is calculated as 1.0), and ratio of maximum to minimum opening diameter; Distribution characteristics of glandular duct openings.

INTERVENTIONS:
Procedure: The tubular adenoma group — Biopsy or removal of polyps for pathological examination. Collect baseline data such as gender, age, BMI, etc. If the pathology confirms a pure tubular adenoma, the observed object will be included in the group for final comparative analysis.
  Other Names: the colonic innominate groove group
  Groups: The tubular adenoma group

SUMMARY:
This study is to analyze the characteristics of the IIIL opening of the duct in tubular adenoma and the colonic innominate groove under EC endoscopy, in order to improve the ability to tell lesions and the colonic innominate groove under EC endoscopy (Endocytoscopy).

DETAILED DESCRIPTION:
This is a prospective cohort study. The recruitment time for all participants will be 4 months. The tubular adenoma group and the colonic innominate groove group will be paired in a 1:2 ratio, with 32 lesions of tubular adenoma and 64 adjacent innominate groove. It is expected that there will be 32 cases and a total of 96 observation subjects. Analyze and compare the characteristics of the opening of the IIIL duct in tubular adenomas and the colonic innominate groove under EC endoscopy, in order to summarize and differentiate them.

ELIGIBILITY:
Inclusion Criteria:

* Cases of colorectal polyps discovered in our hospital and undergoing EC endoscopic examination.

Exclusion Criteria:

* 1.Suffering from hereditary polyposis or inflammatory bowel disease, severe intestinal inflammation, or difficulty recognizing normal intestinal mucosa;

  2. History of methylene blue allergy;

  3. Patients who have participated or are currently participating in other clinical trials within the first 4 weeks of enrollment;

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cases of colorectal polyps discovered in our hospital and undergoing EC endoscopic examination.
Sampling Method: Probability Sample
Enrollment: 96 (Estimated)
Dates: Start 2024-03-26 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of opening length to field of view | 10 minutes after the observation of Endocytoscopy
  (more than 1 field of view is calculated as 1.0)

SECONDARY OUTCOMES:
Observation of anatomical location | 10 minutes after the observation of Endocytoscopy
  The anatomical site (ileocecal region, ascending colon, hepatic flexure, transverse colon, Colonic splenic region, descending colon, sigmoid colon, rectum)

OTHER OUTCOMES:
Morphology of IIIL type glandular opening and unnamed sulcus opening | 10 minutes after the observation of Endocytoscopy
  Morphology of IIIL type glandular opening and unnamed sulcus opening after methylene blue staining.Linear or circular pit pattern.
Distribution characteristics of glandular opening | 10 minutes after the observation of Endocytoscopy
  Magnified to the maximum magnification of EC endoscopy to the clearest cell level (approximately 520 times), and observed the morphology of the opening of the IIIL type glandular duct and the opening of the colonic innominate groove, including the morphology of cell cytoplasm and nucleus, and distribution characteristics of glandular duct openings. Regular or irregular？

CONTACTS AND LOCATIONS:
Locations (1):
- the First Hospital of Jilin University, Changchun, Jilin, China

IPD SHARING:
Plan to Share IPD: No